CLINICAL TRIAL: NCT00201214
Title: Phase I/II Clinical Trial to Determine the Pharmacokinetics and Safety Profile of Citrulline in Children Undergoing Cardiopulmonary Bypass
Brief Title: Citrulline for Children Undergoing Cardiopulmonary Bypass Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rick Barr, Pediatric Critical Care Faculty, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 281; R01HL073317 (NIH); NCT00178815 (obsolete NCT alias)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Defects, Congenital | interventions — Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Citrulline — Phase I - 150mg/kg IV bolus after initiation of cardiopulmonary bypass with dosage escalation study 50mg/kg, 100mg/kg, 150mg/kg IV at 6, 12, 24, 48 hours post operative. Phase II - 150mg/kg IV bolus after initiation of cardiopulmonary bypass with 9mg/kg/hr continuous IV starting 4 hours post bolus and infusing for 48 hours or discharge from PCCU.

SUMMARY:
This study will determine the pharmacokinetics and safety of intravenous citrulline given to children undergoing cardiopulmonary bypass for the correction of congenital heart defects.

DETAILED DESCRIPTION:
BACKGROUND:

Increased pulmonary vascular tone (PVT) can complicate the postoperative course of the following six surgical procedures for congenital heart defects: 1) unrestrictive ventricular septal defect (VSD) repair; 2) atrioventricular septal (AVSD) repair; 3) arterial switch procedure for transposition of the great arteries (TGA); 4) Norwood I procedure; 5) bidirectional Glenn shunt procedure; and 6) Fontan procedure for single ventricle lesions. PVT is partially controlled by nitric oxide (NO). Arginine, the precursor to NO, is a product of the urea cycle. Preliminary data have been presented regarding 169 infants and children who have undergone one of the six previous surgical procedures. It was found that urea cycle function and plasma arginine levels were significantly decreased in all patients. Furthermore, patients with increased PVT had significantly lower arginine levels compared to patients with normal PVT. Finally, a genetic single nucleotide polymorphism (SNP) in the rate limiting urea cycle enzyme (carbamyl phosphate synthetase I [CPSl T1405N]) appeared to affect postoperative plasma arginine levels and PVT. The hypothesis is that genetic polymorphisms in the rate limiting urea cycle enzyme CPSl, and other important enzymes in the urea cycle, influence the availability of NO precursors. It is further hypothesized that perioperative enhancement of urea cycle function with the key urea cycle intermediate (citrulline) will increase plasma arginine and NO metabolites, and prevent elevations in PVT.

DESIGN NARRATIVE:

This phase I/II study will determine the pharmacokinetics and safety of three doses of intravenous citrulline that will be given to children undergoing cardiopulmonary bypass for the correction of congenital heart defects.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiopulmonary bypass via one of the following surgical procedures:

  1. AVSD repair
  2. VSD repair
  3. Bidirectional Glenn
  4. Modified Fontan
  5. Arterial Switch
* Parents willing and able to sign consent

Exclusion Criteria:

* Pulmonary artery or vein abnormalities not being addressed surgically
* Preoperative requirement for mechanical ventilation or intravenous inotrope support
* Any condition that might interfere with study objectives

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2003-12; Primary Completion 2006-01 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Oxygen index (OI) data to assess increased PVT | Measured through the use of continuous mean arterial pressure monitoring
Qp:Qs ratios to assess increased PVT | Measured by blood gases collected 48 hours post-operative
Increased PVT as measured by a sustained mean pulmonary artery pressure greater than 20 mm Hg for at least 2 hours during the first 24 hours postoperatively | Measured through the use of continuous mean arterial pressure monitoring 48 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Frederick E. Barr, MD, MSCI, Study Chair — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768